CLINICAL TRIAL: NCT02541266
Title: Imaging in Clinical Trials - a Questionnaire Study to Assess Impact of Imaging Regimes on Patient Participation
Acronym: ASK
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: 15 LO 1189
Record Dates: First submitted 2015-07-22; First posted 2015-09-04 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: Imaging; Questionnaire
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Patients currently recruited to studies with imaging at The Marsden
  Interventions: Other: Questionnaire
- Group 2: Patients who have previously participated in studies with imaging at The Marsden
  Interventions: Other: Questionnaire
- Group 3: Patients attending for scans as part of their clinical pathway
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A short questionnaire (9 questions) will be given to the participants to complete.

SUMMARY:
This research is aimed at finding out what may influence the decision of patients to participate in trials involving imaging so that the investigators may improve our future studies so they are more patient focused and acceptable in regards to scan schedules.

DETAILED DESCRIPTION:
This is a questionnaire study aimed at gaining a greater understanding of the patient perspective on undertaking imaging procedures, MRI and PET/CT, for research purposes. The study is to evaluate the patient opinion and perceptions of the burden of imaging associated with research. We will look at different scanning procedures of varying duration, intensity, frequency and scheduling; this will enable us to have a better understand of the factors that influence participation in research and thus help us develop protocols that are more patient focused and acceptable.

ELIGIBILITY:
Inclusion Criteria

* Being treated at The Royal Marsden Hospital
* Over the age of 18
* Having imaging (MRI or PET/CT) as part of research or clinical care.
* Group 1

  * Currently enrolled in a research project that involves imaging (either MRI or PET/CT)
* Group 2

  * Previously enrolled in a research project that involved imaging (either MRI or PET/CT), where the patients involvement in the research project has now ended.
* Group 3

  * Patients attending the MRI or PET/CT departments for imaging as part of their standard clinical care.

Exclusion Criteria -

* Inability to complete the questionnaire.
* Previously completed questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients recruited to studies with imaging Group 2: Patients who have previously participated in studies with imaging Group 3: Patients attending for scans as part of their clinical pathway
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-04-01; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Factors that affect patient participation in imaging research | Duration of Study - 1 year
  Factors about an imaging scan - type, length, frequency or scheduling (timing in relation to treatment) - that are perceived as a significant burden when considering participation in a research study involving imaging.

SECONDARY OUTCOMES:
Factors affecting participation in the different patient categories | Duration of Study - 1 year
Effect of current participation in a study on the perceived acceptability of imaging burden | Duration of Study - 1 year
Do opinions change after undergoing imaging procedures | Duration of Study - 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom